CLINICAL TRIAL: NCT03190005
Title: Downstream Molecular Signals of P2Y12 Receptors in Hyporeactive Patients Under Clopidogrel Treatment (A Possible Mechanism of HOTPR:High On- Treatment Platelet Reactivity)
Brief Title: Downstream Molecular Signals of P2Y12 Receptors in Hyporeactive Patients Under Clopidogrel Treatment A Possible Mechanism of HOTPR(High On-Treatment Platelet Reactivity)
Status: Completed | Type: Observational
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Yueh-Chung, Chen, Principal Investigator, Taipei City Hospital
Other Study IDs: TCHIRB-10603117-E
Record Dates: First submitted 2017-06-06; First posted 2017-06-16 (Actual); Results first posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2017-06

CONDITIONS: Stable Angina
Keywords: PRU; P2Y12 receptor
MeSH Terms: conditions — Angina, Stable | interventions — Clopidogrel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — downstream molecular signals of P2Y12 receptor in the platelet(Platelet Rich Plasma).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- group 1: placebo control without medication.
  Interventions: Drug: Placebos
- group 2: hyper-reactive responser after clopidogrel.
  Interventions: Drug: clopidogrel
- group 3: hypo-reactive responser after clopidogrel.
  Interventions: Drug: clopidogrel
- group 4: normo-reactive responser after clopidogrel.
  Interventions: Drug: clopidogrel
- group 5: reaction after OPC-13013
  Interventions: Drug: clopidogrel
- group 6: reaction after AR-C
  Interventions: Drug: clopidogrel
- group 7: reaction after simastatin
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: clopidogrel — routine Dual antiplatelet therapy after stent implantation, then check PRU(platelet reactivity unit)
  Groups: group 2; group 3; group 4; group 5; group 6; group 7
Drug: Placebos — no medication, healthy subjects.
  Groups: group 1

SUMMARY:
The investigators designed the following experiment to observe the pattern of administration in vitro, which can be completely excluded liver enzyme cytochrome P450 metabolism under the influence and observe the relevant P2Y12 receptor downstream signal changes, hope in the above experiments, that the human body directly for the difference between the existence of drug reactions exist.

DETAILED DESCRIPTION:
Platelet reactivity has been accepted as an indicator of the reaction of the P2Y12 inhibitor during treatment, currently, the existing evidence to support the post-treatment platelet activity can be used to distinguish the potential risk among patients who received percutaneous transluminal coronary angioplasty after ischemic / thrombotic events. The risks of stent thrombosis, of which, by analysis of the PRU (P2Y12 reaction units) value level of VerifyNow System has been considered an international standard tools. PRU value by VerifyNow system can easily and quickly showed platelet reactivity relative to short or long term risk stratification under dual antiplatelet agents(aspirin and clopidogrel) after stents implantation. High PRU response units (drug poor responders) in accordance with the 2013 publication of the European Society of Cardiology guidelines defined of platelet function, is PRU not less than 208(≥208).

The investigators ran a previous related plan within 2014 under the medical study project budget of the Taipei City hospital, which named "platelet reactivity as a post-percutaneous coronary stent implantation antiplatelet adjust the reference", it has been figured that responsibility under the P2Y12 receptor inhibitors were significantly different between the taiwanese and Caucasians (taiwanese revealed clopidogrel lower responsive, but stronger reaction to ticagrelor), although "low" response to clopidogrel between taiwanese (In fact, according to our experiments, 30 days after medication, the rate of HOTPR-High On- Treatment Platelet Reactivity; namely PRU≥208, the taiwanese and Caucasians are very close to each), but it has relative lower subacute stent thrombosis rate than the Caucasian at 30 days(This reaction is also known as the "Asian paradox" ), according to literature known abroad because of the high prevalence of CYP2C19 point gene deletion rate among the Asians (compare with Caucasians: ~ 65% vs ~ 30%); there also suggested other possible explanations: Caucasian factor V Leiden (G1691A) and prothrombin (G20210A) a higher proportion of mutations, on hemostatic factors (fibrinogen, d-dimer, and factor VIII) and plasma endothelial activation markers (such as von Willebrand factor, intercellular adhesion molecule 1, and E-selectin) existed differences between the races; in addition, a number of different indicators of inflammation, such as CRP. Asians show lower level CRP than the Caucasians. However, did the investigators found the true answer? So, the investigators designed the following experiment, through the mode of drug administration in vitro, can completely exclude the influence of the liver metabolic enzyme cytochrome P450, and observe the relevant downstream signals of P2Y12 receptors. The investigators believed through the current study, the internal differences in drug responsibility can be clarified.

ELIGIBILITY:
Inclusion Criteria:

* DAPT(Dual antiplatelet therapy) after regular stent implantation.

Exclusion Criteria:

* allergy to DAPT(Dual antiplatelet therapy). major bleeding intolerance to DAPT(Dual antiplatelet therapy).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: stable angina who received routine dual antiplatelet agents therapy.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei city hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Started | 5 | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: patient receive different anti-platelet drug(in vivo or in vitro)
Units Other Than Participants: blood samples
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 35
Number analyzed (blood samples) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 3 | 2 | 2 | 3 | 3 | 20
  >=65 years | 2 | 1 | 2 | 3 | 3 | 2 | 2 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.52 (11.12) | 64.92 (13.24) | 66.89 (10.72) | 63.35 (13.62) | 65.09 (11.13) | 61.23 (10.34) | 68.32 (15.12) | 67.36 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 2 | 2 | 1 | 2 | 13
  Male | 3 | 2 | 4 | 3 | 3 | 4 | 3 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: PRU(Platelet Rreactivity Unit) 24 Hours After DAPT(Dual AntiPlatelet Therapy) Western Blot After Medication
Description: PRU(Platelet Rreactivity Unit) 24 hours after DAPT(Dual AntiPlatelet Therapy) Western blot after medication
Time Frame: 24 hours
Population: PRU(Platelet Rreactivity Unit) 24 hours after DAPT(Dual AntiPlatelet Therapy) Western blot after medication
Measure: Mean (Standard Deviation); unit: PRU(Platelet Rreactivity Unit)
Units Other Than Participants: blood sample
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5
Number analyzed (blood sample) | 5 | 5 | 5 | 5 | 5 | 5 | 5
PRU(Platelet Rreactivity Unit) | 148 (3) | 289 (4) | 79 (1) | 132 (6) | 81 (3) | 62 (2) | 114 (9)

ADVERSE EVENTS:
Time Frame: 1 year
Description: major/minor drug reaction
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT03190005/SAP_000.pdf
  • Informed Consent Form (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT03190005/ICF_001.pdf
  • Study Protocol (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT03190005/Prot_002.pdf